CLINICAL TRIAL: NCT00000938
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial of the Safety and Efficacy of Ceftriaxone and Doxycycline in the Treatment of Patients With Seronegative Chronic Lyme Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMID 97-003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease | interventions — Ceftriaxone; Doxycycline

INTERVENTIONS:
Drug: ceftriaxone
Drug: doxycycline

SUMMARY:
Lyme disease is the most common tick-borne disease in the United States. It is caused by the spirochete Borrelia burgdorferi. It may exist in a chronic form and be the result of: 1) persistent infection by B. burgdorferi; 2) damage caused by the original infectious process; or 3) the presence of coinfection with another organism transmitted by Ixodes ticks. The purpose of this study is to determine the safety and effectiveness, in seronegative patients, of intensive antibiotic treatment in eliminating symptoms of Chronic Lyme Disease (CLD).

DETAILED DESCRIPTION:
Sixty-six patients will be enrolled in this study. Each patient will be assigned to one of two groups and will be randomly selected to receive either antibiotic therapy or placebo; but, the assignment of medication will not be made known to the patient or administering doctor. Antibiotic or placebo will be given intravenously (IV) for 30 consecutive days and then orally for the next 60 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Are at least 18 years of age.
* Are seronegative for antibodies against B. burgdorferi antigens by Western Blot at enrollment.
* Have documented history of acute Lyme disease.
* Have had a rash (erythema migrans) that resembles a bullseye. This skin aberration usually occurs after a tick bite in late spring, summer, or early fall and is sometimes accompanied by fatigue, fever, headache, mild stiff neck, arthralgia or myalgia.
* Have had one or more clinical features typical of Lyme disease acquired in the United States (see technical summary)
* Have had one or more of the following symptoms and conditions that have persisted for at least 6 months (but less than 12 years) and are not attributable to another cause or condition: a) widespread musculoskeletal pain and fatigue that began coincident with or within 6 months following initial infection with B. burgdorferi. b) certain neurologic symptoms including memory impairment and nerve pain, beginning within 6 months following initial infection with B. burgdorferi.
* Have had a physician-documented history of prior antibiotic treatment with a currently recommended antibiotic regimen.

Exclusion Criteria:

You will not be eligible for this study if you:

* Have previously enrolled in this study.
* Are pregnant, lactating, or unable to use birth control measures during the treatment period of this study.
* Are taking chronic medication that could interfere with evaluation of symptoms.
* Are taking or have taken various medications that could interfere with the evaluation of symptoms (see technical summary).
* Are hypersensitive to ceftriaxone or doxycycline.
* Have active inflammatory synovitis.
* Have another disease that could account for symptoms of acute Lyme disease.
* Have another serious or active infection.
* Are unable to tolerate an IV.
* Have tested positive for Borrelia DNA in plasma or cerebrospinal fluid at the time of initial evaluation for study.
* Have tested seropositive by Western Blot (these patients may be offered enrollment in seropositive study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Mark Klempner, Boston, Massachusetts, United States